CLINICAL TRIAL: NCT06461091
Title: A Prospective, Single-arm, Exploratory Clinical Study of the Efficacy and Safety of Total Myeloid Irradiation (TMI) in the Treatment of Adult Acute Lymphoblastic Leukemia
Brief Title: the Efficacy and Safety of Total Myeloid Irradiation (TMI) in the Treatment of Adult Acute Lymphoblastic Leukemia
Acronym: TMI
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2024023
Record Dates: First submitted 2024-05-13; First posted 2024-06-14 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-05

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: TMI — Observing the efficacy and safety of allogeneic hematopoietic stem cell transplantation in treating adult acute lymphoblastic leukemia with a conditioning regimen including total marrow irradiation (TMI) in individuals aged 16 years and older: Primary Exploratory Endpoint: Event-free survival at 1 year post allogeneic hematopoietic stem cell transplantation (EFS).

SUMMARY:
Observation of event-free survival, engraftment rate, overall survival (OS), and safety data in patients aged ≥16 years with acute lymphoblastic leukemia (ALL) receiving a conditioning regimen including total marrow irradiation (TMI) followed by allogeneic hematopoietic stem cell transplantation. Aim to further enhance transplant outcomes in ALL patients based on the existing basis.

DETAILED DESCRIPTION:
Observation of event-free survival, engraftment rate, overall survival (OS), and safety data in patients aged ≥16 years with acute lymphoblastic leukemia (ALL) receiving a conditioning regimen including total marrow irradiation (TMI) followed by allogeneic hematopoietic stem cell transplantation. Aim to further enhance transplant outcomes in ALL patients based on the existing basis.Exploratory Endpoint: Event-free survival at 1 year post allogeneic hematopoietic stem cell transplantation (EFS).Secondary Exploratory Endpoints: (1) Rate of granulocyte and platelet hematopoietic recovery. (2) Incidence of toxicity related to the conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for inclusion in this study must meet all of the following criteria: (1) Definitive diagnosis of acute lymphoblastic leukemia requiring allogeneic hematopoietic stem cell transplantation. (2) Age greater than or equal to 16 years.

Exclusion Criteria:

* Subjects meeting any of the following criteria are not eligible for inclusion in this study: (1) Patients with extramedullary infiltration (excluding central nervous system leukemia). (2) Patients undergoing second transplantation. (3) Patients with concurrent malignancies. (4) Patients with malignancies secondary to a second tumor. (5) Patients assessed by the investigator to have accompanying diseases that are deemed to pose a serious risk to the patient's life or interfere with the patient's completion of this study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients（ aged ≥16 years） with acute lymphoblastic leukemia (ALL) paining to receive allogeneic hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Event-free survival at 1 year post allogeneic hematopoietic stem cell transplantation (EFS). | 1YEAR
  Event-free survival at 1 year post allogeneic hematopoietic stem cell transplantation (EFS).

SECONDARY OUTCOMES:
(1) Rate of granulocyte and platelet hematopoietic recovery. | 1YEAR
  (1) Rate of granulocyte and platelet hematopoietic recovery.
(2) Incidence of toxicity related to the conditioning regimen. | 1YEAR
  (2) Incidence of toxicity related to the conditioning regimen.

IPD SHARING:
Plan to Share IPD: No